CLINICAL TRIAL: NCT00042887
Title: Chemoresection With 4 Weekly Intravesical Instillations Of Mitomycin C Versus Transurethral Resection (TUR) Followed By One Single Immediate Instillation Of Mitomycin C In Single, Small, Papillary Stage Ta, T1 Bladder Tumors: A Prospective Randomized Phase III Trial
Brief Title: Chemotherapy With or Without Surgery in Treating Patients With Bladder Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-30004; EORTC-30004
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer; recurrent bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Mitomycin

INTERVENTIONS:
Drug: mitomycin C
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Infusing chemotherapy drugs directly into the bladder may kill more cancer cells. It is not yet known if surgery followed by chemotherapy is more effective than chemotherapy alone in treating bladder cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy alone with that of transurethral resection followed by chemotherapy in treating patients who have bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of chemoresection with 4 weekly intravesical instillations of mitomycin vs transurethral resection followed by 1 instillation of mitomycin in patients with low-risk superficial transitional cell carcinoma of the bladder.
* Compare the disease-free survival of patients treated with these regimens.
* Determine the response rate at 6 weeks in patients treated with chemoresection.
* Determine the percent of patients with tumor at 6 weeks treated with transurethral resection.
* Compare the quality of life of patients treated with these regimens.
* Compare the side effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease status (primary vs recurrent) and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo chemoresection with intravesical instillation of mitomycin once weekly for 4 weeks.
* Arm II: Patients undergo transurethral resection followed within 1-6 hours by intravesical instillation of mitomycin.

Quality of life is assessed at baseline, at week 1 (arm II only), at week 5 (arm I only), and then at week 6.

Patients are followed at weeks 6 and 19, every 6 months for 3 years, and then annually for 2 years.

PROJECTED ACCRUAL: A total of 1,000 patients (500 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically confirmed solitary primary or recurrent papillary transitional cell carcinoma of the bladder

  * Ta or T1
* Tumor no greater than 2 cm in diameter
* Negative urine cytology
* No suspicious lesions in bladder requiring biopsy
* No tumors in the prostatic urethra or upper urinary tract
* No prior history of T1 G3 tumors, muscle invasive tumors (T2 or greater), or carcinoma in situ

PATIENT CHARACTERISTICS:

Age

* 80 and under

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* HIV negative
* No active intractable or uncontrollable bladder infection
* No urethral strictures that would preclude endoscopic procedures or repeated catheterization
* No prior or concurrent congenital or acquired immune deficiency syndrome
* No other prior or concurrent malignancy except cured basal cell skin cancer or intraepithelial cancer of the cervix
* No prior or concurrent leukemia or Hodgkin's disease
* No concurrent disease for which general anesthesia is contraindicated
* No psychological, familial, sociological, or geographical condition that would preclude study compliance
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 12 months since prior BCG vaccine

Chemotherapy

* At least 1 year since prior mitomycin

Endocrine therapy

* Not specified

Radiotherapy

* No prior pelvic radiotherapy

Surgery

* No prior organ transplant

Other

* At least 3 months since prior intravesical treatment

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2002-05; Primary Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willem Oosterlinck, MD, PhD, Study Chair — University Ghent
Locations (12):
- Belgium (4):
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Virga Jesse Hospital, Hasselt
  - U.Z. Gasthuisberg, Leuven
- Italy (2):
  - Universita Di Palermo, Palermo
  - Ospedale S.S. Annunziata, Savigliano
- Netherlands (4):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Jeroen Bosch Ziekenhuis, NL'S Hertogenbosch
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
- Comenius University School of Medicine, Martin, Slovakia
- Dokuz Eylul University School of Medicine, Izmir, Turkey (Türkiye)